CLINICAL TRIAL: NCT00162825
Title: Role of CD7 in Skin Inflammation and Psoriasis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261700717
Record Dates: First submitted 2005-09-12; First posted 2005-09-13 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2003-06

CONDITIONS: Psoriasis; Inflammation
Keywords: Psoriasis, T cell, inflammation, CD7, cytokine
MeSH Terms: conditions — Psoriasis; Inflammation

SUMMARY:
Role of CD7 in skin inflammation and psoriasis

DETAILED DESCRIPTION:
Psoriasis is a debilitating, chronic inflammatory skin disorder characterized by scaly skin patches caused by infiltration of inflammatory cells into the dermis and epidermis, with secondary epidermal cell (keratinocyte) hyperproliferation. Psoriasis is a complex disease and a combination of genetic and environmental factors are likely to be causative. T-cell-mediated immune process, including cytokines (eg. IFN-γ) and chemokines, play an essential role in psoriasis. Susceptibility genes for psoriasis map to PSORS1 in the HLA region at chromosome 6p21, PSORS2 in the chromosome 17q24-q25, and others.

Recently our colleagues in the Academia Sinica and we performed a genome-wide linkage analysis with polymorphic microsatellites in one five-generation affected psoriasis kindred, and the result revealed a close linkage at D17S928, close to CD7. CD7+ T cells produce IFN-γ when activated, and have been located in skin inflammatory lesions. Therefore, in this study we first want to examine the role of CD7 in skin inflammations conditions. CD7+ cells will be stimulated by a variety of methods, and will be used to treat keratinocyte cultures or be injected intradermally to mice. We will watch for skin inflammation and possible proliferation and changes in keratinocytes. Possible changes in CD7 function in patients with psoriasis will be explored, for example, polymorphisms of the CD7 gene may predispose skin inflammation and abnormal interaction with the keratinocytes. CD7- T cells, which could be derived from CD7+ cells and are enriched in skin inflammation lesions, secrete the Th2 cytokine IL-5. We are also interested in the mechanism and the consequences of this CD7 shift. We hope this study will be helpful in the understanding and management of skin inflammation conditions, including psoriasis.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of psoriasis

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-01; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: whu-Liang Hwu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan